CLINICAL TRIAL: NCT00295893
Title: Randomized Phase II Study of Docetaxel, Adriamycin, and Cytoxan (TAC) Versus Adriamycin/Cytoxan, Followed by Abraxane/Carboplatin (ACAC) +/- Trastuzumab as Neoadjuvant Therapy for Patients With Stage II-III Breast Cancer
Brief Title: Combination Chemotherapy With or Without Trastuzumab in Treating Patients With Stage II or Stage III Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05015; P30CA033572 (NIH); CDR0000455631 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer; Paget disease of the breast with invasive ductal carcinoma; invasive ductal breast carcinoma with predominant intraductal component; invasive ductal breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; comedo ductal breast carcinoma; invasive lobular breast carcinoma with predominant in situ component; invasive lobular breast carcinoma; mucinous ductal breast carcinoma; papillary ductal breast carcinoma; tubular ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Breast Neoplasms, Male; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; Trastuzumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide (Active Comparator): Patients receive doxorubicin hydrochloride IV, cyclophosphamide IV, and docetaxel IV on day 1. Treatment repeats every 21 days for 6 courses.
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride
- Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin (Experimental): Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1; treatment repeats every 2 weeks for 4 courses. Patients then receive carboplatin IV on day 1 and paclitaxel IV on days 1, 8, and 15; treatment with carboplatin and paclitaxel repeats every 4 weeks for 3 courses.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: Carboplatin; Drug: Paclitaxel
- Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and trastuzumab (Experimental): Patients receive chemotherapy as in arm II. They also receive trastuzumab (Herceptin®) IV weekly, beginning with the first doses of paclitaxel and carboplatin.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Biological: Trastuzumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
Drug: docetaxel — Given IV
  Arms: Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide
Drug: doxorubicin hydrochloride — Given IV
Biological: Trastuzumab — Given IV
  Arms: Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and trastuzumab
Drug: Carboplatin — Given IV
  Arms: Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin; Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and trastuzumab
Drug: Paclitaxel — Given IV
  Arms: Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin; Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and trastuzumab

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy with or without trastuzumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether combination chemotherapy is more effective with or without trastuzumab in treating breast cancer.

PURPOSE: This randomized phase II trial is comparing two different regimens of combination chemotherapy given together with or without trastuzumab to see how well they work in treating patients with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare 2 neoadjuvant chemotherapy regimens (docetaxel, doxorubicin hydrochloride, and cyclophosphamide [TAC] vs doxorubicin and cyclophosphamide followed by paclitaxel and carboplatin [ACAC]), in terms of toxicities and effectiveness as defined by the pathological complete remission rate, in patients with non HER2/neu overexpressing stage II or III breast cancer.
* Evaluate the probability of achieving a pathological complete remission when adding trastuzumab (Herceptin®) to ACAC in the subset of patients with HER2/neu overexpressing stage II or III breast cancer.

Secondary

* Identify prognostic and predictive markers of outcome, recurrence, and targets of therapy.

OUTLINE: This is a randomized study. Patients with non HER2/neu overexpressing tumors are randomized to 1 of 2 treatment arms. Patients with HER2/neu overexpressing tumors are assigned to arm III.

* Arm I: Patients receive doxorubicin hydrochloride IV, cyclophosphamide IV, and docetaxel IV on day 1. Treatment repeats every 21 days for 6 courses.
* Arm II: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1; treatment repeats every 2 weeks for 4 courses. Patients then receive carboplatin IV on day 1 and paclitaxel IV on days 1, 8, and 15; treatment with carboplatin and paclitaxel repeats every 4 weeks for 3 courses.
* Arm III: Patients receive chemotherapy as in arm II. They also receive trastuzumab (Herceptin®) IV weekly, beginning with the first doses of paclitaxel and carboplatin.

Within 4 weeks after completion of chemotherapy with or without trastuzumab (Herceptin®), all patients undergo surgery.

PROJECTED ACCRUAL: A total of 105 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven infiltrating ductal or lobular breast carcinoma

  * Stage II or III disease
  * Inflammatory breast cancer allowed
* Hormone-receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status < 2
* Male or female
* Menopausal status not specified (for female patients)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal (except for patient's with Gilbert's disease)
* Creatinine ≤ 1.2 mg/dL
* Creatinine clearance ≥ 70 mL/min
* Ejection fraction ≥ 50% on MUGA
* No neuropathy ≥ grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No prior malignant disease within the past 5 years, excluding:

  * Squamous cell or basal cell skin carcinoma
  * Stage I or in situ cervical carcinoma
* No noninvasive (in situ) breast carcinoma within the past 5 years

PRIOR CONCURRENT THERAPY:

* At least 5 years since prior antiestrogen treatment for any indication other than breast cancer prevention (tamoxifen, raloxifene, or an aromatase inhibitor)
* No prior radiotherapy to the chest wall

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-09-27 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2026-08-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide: Patients receive 50mg/m2 doxorubicin hydrochloride IV, 500 mg/m2 cyclophosphamide IV, and 75 mg/m2 docetaxel IV on day 1. Treatment repeats every 21 days for 6 courses.
- Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin: Patients receive 60 mg/m2 doxorubicin hydrochloride IV and 600 mg/m2 cyclophosphamide IV on day 1; treatment repeats every 2 weeks for 4 courses. Patients then receive AUC 2 carboplatin IV on day 1 and 100 mg/m2 paclitaxel IV on days 1, 8, and 15; treatment with carboplatin and paclitaxel repeats every 4 weeks for 3 courses.
- Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab: Patients receive chemotherapy as in arm II. They also receive 2 mg/kg trastuzumab (Herceptin®) IV weekly, beginning with the first doses of paclitaxel and carboplatin.
Period: Overall Study
Arm/Group | Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab
Started | 37 | 40 | 44
Completed | 37 | 40 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide: Patients receive 50 mg/m2 doxorubicin hydrochloride IV, 500 mg/m2 cyclophosphamide IV, and 75 mg/m2 docetaxel IV on day 1. Treatment repeats every 21 days for 6 courses.
- Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin: Patients receive 60 mg/m2 doxorubicin hydrochloride IV and 600 mg/m2 cyclophosphamide IV on day 1; treatment repeats every 2 weeks for 4 courses. Patients then receive AUC 2 carboplatin IV on day 1 and paclitaxel IV on days 1, 8, and 15; treatment with carboplatin and 100 mg/m2 paclitaxel repeats every 4 weeks for 3 courses.
- Total: Total of all reporting groups
Arm/Group | Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab | Total
Number analyzed (Participants) | 37 | 40 | 44 | 121
Age, Continuous [Median (Full Range); unit: years] | 50 [33 to 65] | 49 [31 to 68] | 52 [30 to 70] | 50 [30 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 44 | 121
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 10 | 13
  African American | 1 | 3 | 3 | 7
  White | 19 | 17 | 19 | 55
  Hispanic | 14 | 19 | 12 | 45
Region of Enrollment [Number; unit: participants]
  United States | 37 | 40 | 44 | 121

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients With Pathologic Complete Response (pCR)
Description: pCR was defined as no evidence of residual invasive cancer (or very few scattered tumor cells) in primary tumor and lymph nodes.
Time Frame: At the time of surgery within 4 weeks of the end of chemotherapy, up to 10 months
Measure: Count of Participants; unit: Participants
Groups:
- Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab: Patients receive chemotherapy as in arm II. They also receive 2 mg/m2 trastuzumab (Herceptin®) IV weekly, beginning with the first doses of paclitaxel and carboplatin.
Arm/Group | Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab
Number analyzed (Participants) | 37 | 40 | 44
Participants | 6 | 4 | 22

2. Primary Outcome: Count of Patients With Residual Cancer Burden (RCB) Scores of 0 or 1.
Description: RCB score is determined using information on the size of the tumor and the extent of tumor cells in the breast and axillary lymph nodes after neoadjuvant therapy. The higher the RCB score, the more residual breast cancer there is in the breast and lymph nodes:
  RCB-0 = No residual breast cancer RCB-I = Small amount of residual breast cancer RCB-II = Moderate amount of residual breast cancer RCB-III = Extensive (a lot of) residual breast cancer
Time Frame: At the time of surgery within 4 weeks of the end of chemotherapy, up to 10 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab
Number analyzed (Participants) | 37 | 40 | 44
Participants | 11 | 10 | 28

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 2 years and 7 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab
All-Cause Mortality (participants affected / at risk) | 2/37 | 4/40 | 4/44
Serious Adverse Events (participants affected / at risk) | 8/37 | 5/40 | 8/44
Other Adverse Events (participants affected / at risk) | 37/37 | 40/40 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide (N=37) | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin (N=40) | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab (N=44)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Doxorubicin Hydrochloride, and Cyclophosphamide (N=37) | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel and Carboplatin (N=40) | Doxorubicin Hydrochloride and Cyclophosphamide Followed by Paclitaxel, Carboplatin and Trastuzumab (N=44)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 30 (126) | 39 (177) | 43 (197)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 3 (4)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 3 (5)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 4 (6) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (3) | 0 (0) | 5 (5)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 6 (6) | 6 (7) | 9 (11)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 17 (25) | 22 (60) | 22 (45)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (3) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (4) | 0 (0) | 1 (1)
Ventricular trigeminy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 3 (4)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (2)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 3 (5) | 4 (5) | 1 (1)
Eye disorder (Eye disorders) | 2 (2) | 4 (4) | 3 (4)
Eye pain (Eye disorders) | 1 (2) | 2 (3) | 1 (1)
Flashing vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 4 (5) | 7 (11) | 10 (19)
Watering eyes (Eye disorders) | 6 (8) | 5 (8) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 3 (3) | 7 (14)
Abdominal pain (Gastrointestinal disorders) | 7 (12) | 7 (11) | 14 (22)
Constipation (Gastrointestinal disorders) | 18 (30) | 23 (60) | 35 (78)
Diarrhea (Gastrointestinal disorders) | 19 (31) | 18 (30) | 22 (39)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (3) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 14 (30) | 16 (44) | 26 (71)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 9 (16) | 11 (24) | 22 (47)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (4)
Gastritis (Gastrointestinal disorders) | 4 (6) | 2 (2) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 8 (13) | 13 (22) | 15 (23)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 5 (7) | 3 (8)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (5) | 3 (3) | 8 (12)
Nausea (Gastrointestinal disorders) | 30 (79) | 36 (114) | 40 (153)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 8 (10) | 8 (16)
Peritoneal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 3 (5) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (19) | 18 (28) | 21 (37)
Chest pain (General disorders) | 1 (1) | 2 (2) | 8 (8)
Chills (General disorders) | 8 (8) | 11 (11) | 8 (12)
Edema limbs (General disorders) | 20 (34) | 9 (21) | 18 (36)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 35 (137) | 40 (205) | 43 (244)
Fever (General disorders) | 4 (5) | 8 (9) | 8 (11)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 2 (2)
General symptom (General disorders) | 1 (1) | 3 (4) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 3 (3)
Injection site reaction (General disorders) | 1 (1) | 6 (8) | 8 (15)
Irritability (General disorders) | 2 (2) | 2 (3) | 2 (2)
Localized edema (General disorders) | 4 (4) | 3 (3) | 7 (7)
Pain (General disorders) | 7 (11) | 15 (26) | 21 (45)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (5)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Upper respiratory infection (Infections and infestations) | 2 (3) | 8 (8) | 6 (7)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 3 (3) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Intraoperative hepatobiliary injury - Gallbladder (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intraoperative neurological injury - NERVES: Peripheral sensory NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 25 (62) | 25 (77) | 34 (110)
Alkaline phosphatase increased (Investigations) | 10 (26) | 16 (53) | 20 (68)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 31 (109) | 37 (143) | 37 (145)
Coagulopathy (Investigations) | 0 (0) | 2 (3) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haptoglobin decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Hyperbilirubinemia (Investigations) | 1 (2) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 2 (2) | 3 (4) | 1 (1)
Leukocyte count decreased (Investigations) | 14 (37) | 27 (73) | 30 (86)
Leukopenia (Investigations) | 8 (43) | 8 (24) | 4 (12)
Lymphocyte count decreased (Investigations) | 3 (11) | 12 (32) | 12 (44)
Lymphopenia (Investigations) | 6 (33) | 6 (29) | 5 (15)
Neutrophil count decreased (Investigations) | 19 (73) | 29 (66) | 32 (70)
Platelet count decreased (Investigations) | 18 (57) | 18 (33) | 16 (34)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Weight gain (Investigations) | 6 (15) | 3 (3) | 7 (11)
Weight loss (Investigations) | 6 (11) | 9 (25) | 14 (30)
Anorexia (Metabolism and nutrition disorders) | 6 (10) | 11 (15) | 16 (30)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 4 (5) | 1 (3) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 25 (75) | 15 (47) | 14 (59)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (22) | 5 (17) | 4 (11)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (27) | 5 (14) | 4 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (16) | 2 (2) | 2 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (7) | 2 (3) | 5 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 2 (5) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 5 (12) | 2 (2) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (17) | 3 (9) | 1 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 10 (23) | 7 (19) | 16 (47)
Serum calcium decreased (Metabolism and nutrition disorders) | 5 (5) | 4 (6) | 14 (17)
Serum calcium increased (Metabolism and nutrition disorders) | 6 (12) | 8 (16) | 4 (5)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (7) | 3 (3) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 6 (14) | 15 (36) | 17 (35)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 6 (11) | 5 (8) | 8 (13)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (7) | 6 (7) | 15 (22)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (7) | 3 (4) | 4 (5)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 12 (21) | 16 (27)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (19) | 9 (13) | 22 (38)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 7 (11) | 4 (4) | 6 (8)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 4 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 12 (14) | 12 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9) | 11 (13) | 14 (30)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 8 (11) | 20 (34) | 20 (45)
Headache (Nervous system disorders) | 20 (31) | 23 (43) | 28 (76)
Memory impairment (Nervous system disorders) | 2 (2) | 2 (2) | 5 (6)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 8 (10) | 4 (4) | 9 (18)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 28 (71) | 33 (95) | 40 (109)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Taste alteration (Nervous system disorders) | 12 (18) | 12 (18) | 20 (45)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1) | 6 (7)
Anxiety (Psychiatric disorders) | 15 (16) | 12 (19) | 9 (16)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (5) | 10 (16) | 9 (19)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 14 (21) | 19 (27) | 11 (19)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 4 (4) | 3 (4)
Protein urine positive (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (5) | 4 (4) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 4 (6) | 4 (4) | 2 (6)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 2 (3)
Irregular menstruation (Reproductive system and breast disorders) | 12 (18) | 3 (4) | 4 (8)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 4 (5) | 3 (3) | 2 (4)
Vaginal atresia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 3 (3) | 3 (4) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 2 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 9 (12) | 12 (17)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (21) | 23 (33) | 20 (37)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 11 (23) | 19 (29)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 3 (3)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 7 (7) | 9 (12)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (11) | 7 (9)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (56) | 32 (73) | 33 (77)
Atrophy skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6) | 8 (10) | 10 (16)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (6)
Nail disorder (Skin and subcutaneous tissue disorders) | 12 (17) | 14 (25) | 15 (30)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (8) | 8 (11)
Rash desquamating (Skin and subcutaneous tissue disorders) | 10 (13) | 10 (16) | 13 (24)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 7 (7) | 14 (14) | 6 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (11) | 8 (13) | 4 (12)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 13 (15) | 7 (8) | 11 (20)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 1 (1) | 3 (5)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 22 (51) | 21 (63) | 22 (72)
Hypertension (Vascular disorders) | 4 (6) | 6 (14) | 7 (13)
Hypotension (Vascular disorders) | 4 (9) | 4 (6) | 6 (11)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-03-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT00295893/Prot_SAP_000.pdf